CLINICAL TRIAL: NCT01519102
Title: An Open-label, Randomized Two-way, Cross-over Study to Compare Meal-and-carbohydrate-announcement Strategy Versus Meal-announcement Strategy During Closed-loop Regulation of Glucose Levels in a Morning Meal in Adults With Type-1 Diabetes.
Brief Title: Comparison of Closed-loop Operation After Morning Meal With and Without Carbohydrate Counting
Acronym: CLASS02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: McGill University (Other); Montreal Children's Hospital of the MUHC (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Associate Professor of Medicine, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-02
Record Dates: First submitted 2012-01-24; First posted 2012-01-26 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Type-1 Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHO-independent partial insulin bolus with closed-loop (Active Comparator)
  Interventions: Device: Dual Hormone closed-loop system
- CHO-dependent full insulin bolus combined with closed-loop (Active Comparator)
  Interventions: Device: Dual Hormone closed-loop system

INTERVENTIONS:
Device: Dual Hormone closed-loop system — The closed-loop system is composed of three components: continuous glucose system, insulin infusion pumps that infuses insulin and glucagon and a control algorithm that decides on the infusion rates based on sensor readings.

SUMMARY:
Closed-loop strategy is composed of three components: glucose sensor to read glucose levels, insulin pump to infuse insulin and a dosing mathematical algorithm to decide on the required insulin dosage based on the sensor's readings. A dual-hormone closed-loop system would regulate glucose levels through the infusion of two hormones: insulin and glucagon.

The main goal of this project is to assess whether a dual-hormone closed-loop strategy would alleviate the burden of carbohydrate counting from patients with type 1 diabetes (T1D) without a significant degradation in post-meal glucose control.

Each patient will be admitted twice to a clinical research facility. In one visit, patients will eat a morning meal accompanied with a matching insulin bolus (depending on the carbohydrate content of the meal) and glucose levels will be subsequently regulated using dual-hormone closed-loop system. In the other visit, patients will eat the same meal but will inject only a partial insulin bolus (not depending on carbohydrate content of the meal) and the remaining needed insulin will be delivered based on glucose sensor excursions as part of closed-loop operation. If post-meal glucose levels were indifferent between the two visits, then this would suggest that carbohydrate counting may not be necessary during closed-loop operation as the closed-loop system will give any remaining insulin needed to cover the glucose absorbed from the meal. Twelve subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 and ≤ 65 years of old.
* Clinical diagnosis of type 1 diabetes for at least one year. The diagnosis of type 1 diabetes is based on the investigator's judgment and medical history (e.g. history of acido-ketosis, etc.); C peptide level and antibody determinations are not needed.
* The subject will have been on insulin pump therapy for at least 3 months.
* Last (less than 3 months) HbA1c ≤ 12%.

Exclusion Criteria:

* Clinically significant nephropathy, neuropathy (especially clinically significant gastroparesis) or retinopathy as judged by the investigator.
* Recent (< 3 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
* Pregnancy.
* Severe hypoglycemic episode within two weeks of screening.

  • Medication likely to affect with the interpretation of the results: Prandase, Victoza, Byetta and Symlin
* Known or suspected allergy to the trial products or meal contents.
* Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
* Failure to comply with team's recommendations (e.g. not willing to eat snack, not willing to change pump parameters, etc).
* Unreliable carbohydrate counting
* Problems with venous access

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Incremental area under the curve of plasma glucose concentration as compared to pre-meal glucose value of the postprandial glucose excursions | 0-300min

SECONDARY OUTCOMES:
Percentage of postprandial time of plasma glucose concentrations spent in the high range (above 10.0 mmol/l). | 0-300 min
Mean plasma glucose concentration.
Total insulin delivery
Total glucagon delivery
Plasma glucose concentration and incremental plasma glucose concentration at 2 hours postmeal
Postprandial peak and incremental postprandial peak of plasma glucose concentration
Percentage of time of plasma glucose concentrations spent in target range. Target range is defined to be between 4.0 and 10.0 mmol/l for 150 minutes postmeal and between 4.0 and 8.0 mmol/l afterwards
Percentage of postprandial time of plasma glucose concentrations spent in the low range (below 4.0mmol/l) | 0-300min

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherches Cliniques de Montréal (IRCM), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Haidar A, Farid D, St-Yves A, Messier V, Chen V, Xing D, Brazeau AS, Duval C, Boulet B, Legault L, Rabasa-Lhoret R. Post-breakfast closed-loop glucose control is improved when accompanied with carbohydrate-matching bolus compared to weight-dependent bolus. Diabetes Metab. 2014 Jun;40(3):211-4. doi: 10.1016/j.diabet.2013.12.001. Epub 2014 Mar 19. PMID 24656963